CLINICAL TRIAL: NCT00338039
Title: Induction Cetuximab (IM-C225), Gemcitabine and Oxaliplatin, Followed by Radiotherapy With Concurrent Capecitabine, and Cetuximab, Followed by Maintenance Cetuximab and Gemcitabine for Patients With Locally Advanced Pancreatic Cancer
Brief Title: Induction Cetuximab (IM-C225), Gemcitabine, and Oxaliplatin in Pancreatic Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0983
Record Dates: First submitted 2006-01-27; First posted 2006-06-20 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-02

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Cetuximab; C225; Erbitux; Gemcitabine; Oxaliplatin; Eloxatin; Capecitabine; Xeloda
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cetuximab; Gemcitabine; Oxaliplatin; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy + Chemoradation (Experimental): Systemic chemotherapy followed by chemoradiation in locally advanced pancreatic cancer. Cetuximab 500 mg/m^2 intravenous (IV)/week +/-1 day continued throughout induction chemotherapy, chemoradiation and maintenance chemotherapy. Induction Therapy Gemcitabine 1 gm/m^2 over 100 minutes every 2 weeks +/-1 day for 4 doses; Induction Chemotherapy Oxaliplatin 100 mg/m^2 over 120 minutes every 2 weeks +/-1 day for 4 doses. Capecitabine Chemoradiation (to start 2-3 weeks post completion of oxaliplatin and gemcitabine): 825 mg/m^2 by mouth (PO) twice daily Monday-Friday throughout radiation. Conformal radiation therapy to gross disease, total dose = 50.4 Gy delivered in 28 fractions.
  Interventions: Drug: Cetuximab; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Capecitabine; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cetuximab — 500 mg/m^2 IV/week +/-1 day continued throughout induction chemotherapy, chemoradiation and maintenance chemotherapy.
  Other Names: C225; Erbitux; IMC-C225
Drug: Gemcitabine — Induction Therapy: 1 gm/m^2 over 100 minutes every 2 weeks +/-1 day for 4 doses.
  Chemotherapy Maintenance: 1 gm/m^2/week over 100 minutes weekly for 3 weeks then 1 week off.
  Other Names: Gemzar; Gemcitabine Hydrochloride
Drug: Oxaliplatin — Induction Chemotherapy: 100 mg/m^2 over 120 minutes every 2 weeks +/-1 day for 4 doses.
  Other Names: Eloxatin
Drug: Capecitabine — Chemoradiation (to start 2-3 weeks post completion of oxaliplatin and gemcitabine): 825 mg/m^2 by mouth (PO) twice daily Monday-Friday throughout radiation.
  Other Names: Xeloda
Radiation: Radiotherapy — Conformal radiation therapy to gross disease, total dose = 50.4 Gy delivered in 28 fractions.
  Other Names: XRT

SUMMARY:
The primary objective is to evaluate the efficacy of a combination of cetuximab with systemic chemotherapy followed by chemoradiation in locally advanced pancreatic cancer. The primary endpoint is actuarial one-year survival.

The secondary objectives are:

* To evaluate the local tumor response in patients treated with the above regimen.
* To characterize the safety of the above regimen.

DETAILED DESCRIPTION:
Cetuximab is a drug that blocks epidermal growth factor receptor (EGFR). EGFR may be involved in certain types of cancer. When EGFR is stimulated, a series of chemical reactions starts that results in a tumor being "told" to grow. Cetuximab tries to stop these reactions by blocking EGFR. This may stop tumors from growing. Cetuximab has been shown to increase the effect of chemotherapy and of radiation therapy, both of which will also be given in this study.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete medical history and physical exam. Blood (about 2 tablespoons) and urine will be collected for routine tests. Chest x-rays and computed tomography (CT) scans of the abdomen will be done. Women who are able to have children must have a negative urine pregnancy test.

If you are found to be eligible to take part in this study, you will first receive cetuximab every 2 weeks for 8 weeks (4 doses). Cetuximab will be given every 2 weeks throughout the duration of the study. Cetuximab will be continued during the radiation and capecitabine combination, during the retesting stage and then during the chemotherapy that is given after radiation therapy. Cetuximab infusions will be given over approximately 2 hours. Gemcitabine and oxaliplatin chemotherapy will be given once every 2 weeks (4 doses) for 8 weeks. Both drugs are given through a central line and over about 2 hours. Cetuximab will be given first, followed by gemcitabine, and then followed by oxaliplatin. A CT scan and chest X-ray will be done 2 weeks after the last dose (at Week 10).

As long as the tumor has not grown or spread, you will then receive cetuximab, capecitabine, and radiation therapy together. The Capecitabine will be given by mouth twice a day every day of radiation therapy (5 and 1/2 weeks). Radiation therapy will be given once a day for 5 days in a row. It will be given for 5 and 1/2 weeks or 28 treatments. The radiation will be given from 4 directions and focused on the tumor while you are lying on your back. You will continue to receive cetuximab by vein once every 2 weeks during capecitabine and radiation therapy.

After radiotherapy, you will continue to take cetuximab by vein every 2 weeks. The effect of treatment will be evaluated 5-6 weeks after the completion of radiation therapy and capecitabine. A chest x-ray and CT scans will be performed, and about 2 tablespoons of blood will be drawn for routine testing. As long as the tumor has not grown or spread and the side effects are not too severe, you may continue to receive Cetuximab by vein once every 2 weeks . You will also receive Gemcitabine by vein in the same dose as before for 3 out of every 4 weeks as long as the tumor does not grow and the side effects are not too severe. CT scans and chest x-rays will then be done every 2 months to evaluate the status of the tumor.

During the study, you will have physical exams, including weekly blood tests (about 2 tablespoons) each. The possible development of side effects will be closely monitored and could require extra blood and/or urine samples.

You will be taken off study if your disease gets worse or intolerable side effects occur. You may have surgery if at any time during therapy the tumor can be removed surgically. A separate consent form will be used for that situation.

This is an investigational study. Capecitabine, oxaliplatin, and cetuximab are approved by the FDA for colon cancer but have not been approved by the FDA for pancreatic cancer. Up to 69 patients will take part in this multicenter study. Up to 60 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologic or histologic proof of adenocarcinoma of the pancreas is required prior to treatment. Patients can have tumor originating in any part of the pancreas. Islet cell tumors are not eligible. Only patients with non- metastatic, unresectable disease (AJCC 2002 stage T4 NX M0) are eligible. Computed Tomography (CT) findings of lung, liver, peritoneal metastasis are equivocal, are eligible. Patients who cannot undergo resection because of underlying medical problems are also eligible. Diagnosis of Pancreatic Adenocarcinoma by bile duce brushings are acceptable. Patients with regional nodal disease are eligible.
2. All patients must be staged with a physical exam, chest X-ray (CXR), and contrast-enhanced helical thin-cut abdominal CT. Unresectability is defined by CT criteria: a) evidence of tumor extension to the celiac axis or superior mesenteric (SM) artery, or b) evidence on either CT or angiogram of occlusion of the SM vein or SM/ portal vein confluence. If a tumor does not meet this definition and is found to be unresectable at surgical exploration, then that tumor is considered unresectable.
3. Patients must be 18 years and older. There will be no upper age restriction
4. Karnofsky performance status greater than or equal to 70 are eligible.
5. Patients must either be not of child bearing potential or have a negative urine pregnancy test within 72 hours of treatment. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or they have been postmenopausal for at least 12 months.
6. Women of childbearing potential must agree to practice adequate contraception and to refrain from breast-feeding, as specified in the informed consent. Sexually active males must practice contraception during the study.
7. Bone marrow function: absolute neutrophil count (ANC) >1,500/ul. Platelets >100,000/ul.
8. Renal function: creatinine clearance >30 mL/min (calculated with Cockcroft-Gault equation).
9. Hepatic function: Total bilirubin less than 5mg/dL. If the patient required an endobiliary stent, the bilirubin level must have declined on consecutive measurements indicating adequate biliary decompression; alanine aminotransferase (ALT) less than or equal to 5 times the upper limit of normal.
10. Neurologic function: neuropathy (sensory) < Common Toxicity Criteria (CTC) Grade 2.
11. Patients must sign a study-specific consent form, which is attached to this protocol.

Exclusion Criteria:

1. Patients with a history of prior metastatic cancer.
2. Patients must not have significant infection,i.e., requiring intravenous (IV) antibiotics, or other coexistent medical condition that would preclude protocol therapy.
3. Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with ejection fraction less than <30%.
4. Prior therapy which specifically and directly targets the estimated EGFR pathway.
5. Prior severe infusion reaction (bronchospasm, stridor, urticaria and/or hypotension) to a monoclonal antibody.
6. Any prior history of radiotherapy to the abdomen.
7. History or evidence upon physical examination of central nervous system (CNS) disease (e.g., primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of stroke)
8. Prior unanticipated severe reaction to fluoropyrimidine therapy or known hypersensitivity to 5-fluorouracil.
9. Patients who have had an organ allograft.
10. Patients on Coumadin must be changed to Lovenox at least 1 week prior to starting capecitabine. Low dose (1 mg) Coumadin is allowed.
11. Patients taking Sorivudine or Brivudine A must be off of these drugs for 4 weeks prior to starting capecitabine. Patients taking cimetidine must have this drug discontinued. Ranitidine or a drug from another anti-ulcer class can be substituted for cimetidine if necessary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H. Crane, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas (UT) MD Anderson Cancer Center official website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 15, 2005 to June 29, 2009. All recruitment done at hospital and medical clinics.
Groups:
- Chemotherapy + Chemoradation: Systemic chemotherapy followed by chemoradiation in locally advanced pancreatic cancer. Cetuximab 500 mg/m^2 intravenous (IV)/week +/-1 day continued throughout induction chemotherapy, chemoradiation and maintenance chemotherapy. Induction Therapy Gemcitabine 1 gm/m^2 over 100 minutes every 2 weeks +/-1 day for 4 doses; Induction Chemotherapy Oxaliplatin 100 mg/m^2 over 120 minutes every 2 weeks +/-1 day for 4 doses. Capecitabine Chemoradiation (to start 2-3 weeks post completion of oxaliplatin and gemcitabine): 825 mg/m^2 by mouth (PO) twice daily Monday-Friday throughout radiation. Conformal radiation therapy to gross disease, total dose = 50.4 Grey delivered in 28 fractions.
Period: Overall Study
Arm/Group | Chemotherapy + Chemoradation
Started | 69
Completed | 69
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Chemotherapy + Chemoradation: Systemic chemotherapy followed by chemoradiation in locally advanced pancreatic cancer. Cetuximab 500 mg/m^2 IV/week +/-1 day continued throughout induction chemotherapy, chemoradiation and maintenance chemotherapy. Induction Therapy Gemcitabine 1 gm/m^2 over 100 minutes every 2 weeks +/-1 day for 4 doses; Induction Chemotherapy Oxaliplatin 100 mg/m^2 over 120 minutes every 2 weeks +/-1 day for 4 doses. Capecitabine Chemoradiation (to start 2-3 weeks post completion of oxaliplatin and gemcitabine): 825 mg/m^2 by mouth (PO) twice daily Monday-Friday throughout radiation. Conformal radiation therapy to gross disease, total dose = 50.4 Gy delivered in 28 fractions.
Arm/Group | Chemotherapy + Chemoradation
Number analyzed (Participants) | 69
Age Continuous [Median (Full Range); unit: years] | 62 [39 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate
Description: 1-year, 2-year, and 4-year actuarial overall survival (OS) rates defined as number of participants out of total participants alive at 1, 2 or 4 years post baseline treatment.
Time Frame: 1 to 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy + Chemoradation
Number analyzed (Participants) | 69
percentage of participants
  1-year OS Rate | 66.0
  2-year OS Rate | 25.02
  4-year OS Rate | 11.3

2. Primary Outcome: Median Overall Survival
Description: Median survival is defined as the time of initiation of the first dose of chemotherapy to the date of death.
Time Frame: Baseline to disease progression or death, up to 4 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy + Chemoradation
Number analyzed (Participants) | 69
Months | 19.2 [14.2 to 24.2]

ADVERSE EVENTS:
Time Frame: 4 years and 2 months
Arm/Group | Chemotherapy + Chemoradation
Serious Adverse Events (participants affected / at risk) | 4/69
Other Adverse Events (participants affected / at risk) | 11/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Chemoradation (N=69)
normocytic anemia (Blood and lymphatic system disorders) | 1
dehydration (General disorders) | 1
hyponatremia (Blood and lymphatic system disorders) | 1
allergic reaction during infusion (General disorders) | 1
biliary sepsis (Hepatobiliary disorders) | 1
Sepsis/Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3
Hyperglycemia (Blood and lymphatic system disorders) | 3
Fever (General disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Chemoradation (N=69)
nausea (Gastrointestinal disorders) | 7 — associated with anorexia
diarrhea (Gastrointestinal disorders) | 4
anorexia (Gastrointestinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No